CLINICAL TRIAL: NCT04312425
Title: Comparison of Classic and Modified Rapid Sequence Induction on Prevention of Perioperative Gastric Content Regurgitation in Emergency Surgery Under General Anesthesia
Brief Title: Classic and Modified Rapid Sequence Induction for Prevention of Gastric Content Regurgitation
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-SR-093
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Rapid Sequence Induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group C: General anesthesia was induced with classic rapid sequence induction protocol.
  Interventions: Procedure: Classic rapid sequence induction
- Group M: General anesthesia was induced with modified rapid sequence induction protocol.
  Interventions: Procedure: Modified rapid sequence induction

INTERVENTIONS:
Procedure: Modified rapid sequence induction — Modified RSI was put into use in day shift emergency surgery since March 1, 2018. In this scheme, dorsal elevated position and apneic oxygenation technic are applied. Positive pressure mask ventilation is avoided unless necessary. Sellick's technic is not used in this scheme.
  Groups: Group M
Procedure: Classic rapid sequence induction — In classic RSI scheme, patients are in supine position during induction and intubation. Sellick's technic is applied after sedatives and muscle relaxant are given.
  Groups: Group C

SUMMARY:
Induction of anesthesia induces a loss of protective upper airway reflexes and is associated with gastric content regurgitation. Emergency surgery bears a higher risk of gastric content regurgitation because of full stomach, delayed gastric emptying, intestinal obstruction, stroke or other factors. Rapid sequence induction (RSI) of anesthesia was recommended to minimize the risk of regurgitation and aspiration. Classic RSI scheme mainly includes the use of short-acting sedatives and muscle relaxant, together with a manual pressure to the cricoid cartilage (Sellick maneuver) which aims at compressing the esophagus to avoid regurgitation. Though widely recommended, the scheme has been controversial for years. Our department modified the scheme and put it into use in day shift emergency surgery since March 1, 2018. This retrospective analysis is aimed at comparing the effect of classic and modified rapid sequence induction in prevention of gastric content regurgitation in emergency surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients receive emergency surgery under general anesthesia March 1, 2015 to February 29, 2020
* Eighteen years or older

Exclusion Criteria:

* Trachea intubation status on admission
* Tracheotomy
* Bronchoscope surgery
* General anesthesia with laryngeal mask
* Awake intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receive emergency surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 8601 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of gastric content regurgitation | From entering operation room to endotracheal intubation completed.
  The Electronic Anesthesia Record System files contained the word "aspiration" and/or "gastric content" were extracted and carefully evaluated. The events of gastric content regurgitation on admission or observed during tracheal intubation were recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengnian Ding, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No